CLINICAL TRIAL: NCT06795074
Title: Risk of Recurrent Urethral Stricture After Treatment With Paclitaxel-Coated Dilatation Balloon (Optilume) Compared With Non-coated Dilatation Balloon - a Prospective Randomised Multicentre Study
Brief Title: Risk of Recurrent Urethral Stricture After Treatment With Paclitaxel-Coated Dilatation Balloon (Optilume) Compared With Non-coated Dilatation Balloon
Acronym: RUSTIC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Region Skåne (Unknown); Region Stockholm (Other Government); Region Örebro (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RUSTIC; CIV-24-12-050340 (Other: Swedish Medical Agency)
Record Dates: First submitted 2025-01-24; First posted 2025-01-27 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Urethral Stricture
Keywords: drug-coated dilatation balloon
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Paclitaxel-coated dilatation ballon (Experimental): Dilatation of urethral stricture with paclitaxel-coated balloon
  Interventions: Combination Product: Optilume
- Non-coated dilatation balloon (Active Comparator): Dilatation of urethral stricture with non-coated balloon
  Interventions: Device: UroMax Ultra

INTERVENTIONS:
Combination Product: Optilume — Dilatation with drug-coated balloon
  Arms: Paclitaxel-coated dilatation ballon
Device: UroMax Ultra — Dilatation with non-coated balloon
  Arms: Non-coated dilatation balloon

SUMMARY:
Urethral strictures are often initially treated endoscopically with dilatation or direct visual internal urethrotomy (DVIU), a procedure where the stricture is incised through the vision of a cystoscope. These methods are easy to perform, they are often well tolerated under local anesthesia and they have a low risk of complications. One disadvantage is the relatively low success rate which is 20-60% when used as a first intervention and considerably lower after several interventions. Instead of repeated endoscopic procedures, it is advisable to perform open urethroplasty. Urethroplasty has a success rate of 65-91% but a higher risk of complications and requires general anesthesia. Therefore, there is a need for a treatment option for recurrent urethral strictures after DVIU or dilatation, before the urethroplasty is performed.

Optilume is a CE-marked paclitaxel-coated dilatation balloon used for treatment of urethral strictures. The industry-sponsored randomised ROBUST III trial from 2022 showed a 75% success rate with Optilume but it is not sure if the results can be generalised to patients who would otherwise be candidates for open urethroplasty and whether the drug coating per se increases the efficacy of balloon dilatation. The aim of this study is to investigate whether the addition of paclitaxel-coating can increase the success rate and decrease the need for additional interventions and open urethroplasty for individuals who has a recurrent urethral stricture following at least one previous endoscopic intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Urethral stricture recurrence after at least one internal urethrotomy or dilatation
* Penile or bulbar stricture
* Length of stricture ≤ 2 cm
* Eligible for open urethroplasty
* Able to give informed consent

Exclusion Criteria:

* Stricture of the meatus
* Sclerosis of the bladder neck
* Multiple strictures < 16 Ch
* Complete stricture without any lumen
* Previous dilatation with paclitaxel-coated balloon
* Previous radiation therapy of the pelvis (e.g. for prostate cancer)
* Previous pelvic fracture
* Urethral malignancy
* Presence of urethral fistula
* Presence of urethral condyloma
* Previous open urethroplasty
* Chronic urinary retention secondary to detrusor inactivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Functional recurrent stricture | Within 18 months of treatment
  Recurrence within 18 months of a functional urethral stricture, defined as:
  1. Use of clean intermittent dilatation or
  2. Retreatment with dilatation balloon or internal urethrotomy or
  3. Need for open urethroplasty or other open procedure

SECONDARY OUTCOMES:
Anatomical recurrent stricture | Within 18 months of treatment
  Anatomical recurrent stricture, defined as impassable with a 16 Fr flexible cystoscope
Qmax | At 6 and 18 months after treatment
  Change in maximum urinary flow after treatment
Time micturition | At 6 and 18 months after treatment
  Change in time micturition (seconds for first 1dL voided urine)
Urethral Stricture Score | At 6, 12 and 18 months after treatment
  Patient reported outcome measure (Urethral Stricture Surgery (USS)-PROM). Score from 0-24, higher indicates worse symptoms. Also includes a quality-of-life question and Peeling's voiding picture.

CONTACTS AND LOCATIONS:
Locations (4):
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - Skåne University Hospital, Malmo
  - Örebro University Hospital, Örebro
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No
Not allowed by ethical review authority